CLINICAL TRIAL: NCT00797849
Title: A Randomized, Controlled Study to Evaluate the Effectiveness of Farabloc for Chronic Phantom Limb Pain Among Veteran Amputees
Brief Title: Controlled Study of Farabloc for Chronic Phantom Limb Pain Among Veteran Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Samueli Institute for Information Biology (Other)
Responsible Party: An-Fu Hsiao, M.D., Ph.D., Southern California Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: #871; Contract 1 EA-0000078; Subaward for W81XWH-06-1-0279
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Phantom Limb Pain
Keywords: phantom limb pain; amputees; Farabloc; Phantom limb pain in the missing limb of Veteran amputees
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Wear prosthetics laminated with Farabloc surrounding the liner. If not wearing prosthetics, subject needs to wear Farabloc sock or glove over shrinker.
  Interventions: Device: Farabloc Limb Cover
- 2 (Sham Comparator): Wear prosthetics laminated with sham material surrounding the liner. If not wearing prosthetics, subject needs to wear sock or glove over shrinker.
  Interventions: Device: Sham Limb Cover

INTERVENTIONS:
Device: Farabloc Limb Cover — Wear prosthetics, sock or glove laminated with Farabloc
  Other Names: FARABLOC - LC
  Arms: 1
Device: Sham Limb Cover — Wear prosthetics, sock or glove laminated with sham material
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine if the group using Farabloc shows a greater reduction in pain levels than the group not using Farabloc at 6-week, 12-week and 1-month post treatment follow-ups.

DETAILED DESCRIPTION:
Phantom limb pain (PLP)is a painful sensation perceived in the missing limb after amputation and may be triggered by episodes of stump pain. A growing body of literature indicates that 50-80% of amputees may have PLP. Farabloc cloth is a noninvasive, alternative therapy developed by Farabloc Development Corporation for use by amputees with PLP. The Farabloc Corporation will be donating them to the VA Long Beach for use in this study without charge. Farabloc is a non-toxic and non-invasive treatment with promising preliminary pilot data. Metallic fibers consisting mainly of iron (85.3%) and nickel (10.0%) are woven into a nylon fabric that can be custom made into socks, gloves, limb covers, etc. Farabloc can be laminated into the socket and in the design of the prosthetic without weakening or adding significant weight to it. The exact mechanism of action is unknown for Farabloc, however, it is theorized that the fabric shields high frequency electromagnetic fields that may cause cellular damage and subsequent pain.

Subjects over 18 will be recruited from the VA Long Beach Prosthetic Clinic. Eligible subjects who are interested to participate, will be scheduled for a screening visit. Written informed consent will be obtained before enrollment. Enrolled subjects will be randomly assigned to either the Farabloc or sham Farabloc group. Assignment is double-blind to study participants, prosthetist, Farabloc Corporation and the research assistant throughout the study. Only the project coordinator and PI will know the random assignment.

Farabloc intervention will consist of wearing prosthetics laminated with Farabloc surrounding the liner or, if not wearing prosthetics, subject will wear Farabloc sock or glove over shrinker. Sham intervention will consist of wearing prosthetics laminated with sham fabric surrounding the liner or, if not wearing prosthetics, subject will wear sock or glove made of sham fabric over shrinker. All subjects will receive at least two socks.

Data for PLP pain levels and health-related quality of life will be collected during baseline, 6-week, 12-week and 1-month post treatment follow-up. Research staff will administer these surveys and collect data in person. The amount of health care utilization will be measured 12-week prior ot enrollment and 12-week follow-up. Monitoring adherence to protocol by phone call will be made during the treatment at 3-week and 9-week followup.

Study participants will receive a total of $50 for their participation in this study ($20 for baseline and $10 for each of the three follow-up visits). At the end of the study, participants can choose to keep the active or sham Farabloc. If the true Farabloc turns out to be an effective treatment for phantom limb pain, subjects assigned to the sham Farabloc intervention will b offered the option to be treated with true Farabloc free of charge aftr conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Upper or lower extremity amputees with healed stumps
* Experience episodes or intermittent PLP
* At least 3 episodes of PLP during the previous 6 weeks
* Have not used Farabloc within the last 6 months

Exclusion Criteria:

* Pregnant women are excluded from the study
* Stump complications (e.g., cellulites and stump pain caused by new bone spur within the past 12 months
* Previous use of Farabloc within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be pain as measured by the Numerical Pain Rating Scale (NPRS). | Measurements will be obtained at baseline, and 6-week and 12-week follow-ups

SECONDARY OUTCOMES:
A secondary outcome will measure health-related quality of life using the 36-item Sort Form Health Survey (SF-36). | The assessment will be conducted at pretest, 6-week, 12-week and 1-month post treatment.
Measurement of health care utilization will be conducted by comparing the numbers of outpatient visits emergency room visits and inpatient hospitalizations using the VA electronic medical system CPRS. | At 12-week pretreatment and 12-week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: An-Fu Hsiao, M.D., Ph.D., Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Background] Adams PF, Hendershot GE, Marano MA; Centers for Disease Control and Prevention/National Center for Health Statistics. Current estimates from the National Health Interview Survey, 1996. Vital Health Stat 10. 1999 Oct;(200):1-203. PMID 15782448
- [Background] Ephraim PL, Dillingham TR, Sector M, Pezzin LE, Mackenzie EJ. Epidemiology of limb loss and congenital limb deficiency: a review of the literature. Arch Phys Med Rehabil. 2003 May;84(5):747-61. doi: 10.1016/s0003-9993(02)04932-8. PMID 12736892
- [Background] Potter BK, Scoville CR. Amputation is not isolated: an overview of the US Army Amputee Patient Care Program and associated amputee injuries. J Am Acad Orthop Surg. 2006;14(10 Spec No.):S188-90. doi: 10.5435/00124635-200600001-00041. PMID 17003197
- [Background] Lin DL, Kirk KL, Murphy KP, McHale KA, Doukas WC. Evaluation of orthopaedic injuries in Operation Enduring Freedom. J Orthop Trauma. 2004 May-Jun;18(5):300-5. doi: 10.1097/00005131-200405000-00006. PMID 15105752
- [Background] Islinger RB, Kuklo TR, McHale KA. A review of orthopedic injuries in three recent U.S. military conflicts. Mil Med. 2000 Jun;165(6):463-5. PMID 10870364
- [Background] Korver AJ. Amputees in a hospital of the International Committee of the Red Cross. Injury. 1993 Oct;24(9):607-9. doi: 10.1016/0020-1383(93)90124-o. PMID 8288381
- [Background] Sherman RA. Phantom limb pain. Mechanism-based management. Clin Podiatr Med Surg. 1994 Jan;11(1):85-106. PMID 8124659
- [Background] Ephraim PL, Wegener ST, MacKenzie EJ, Dillingham TR, Pezzin LE. Phantom pain, residual limb pain, and back pain in amputees: results of a national survey. Arch Phys Med Rehabil. 2005 Oct;86(10):1910-9. doi: 10.1016/j.apmr.2005.03.031. PMID 16213230
- [Background] Kooijman CM, Dijkstra PU, Geertzen JHB, Elzinga A, van der Schans CP. Phantom pain and phantom sensations in upper limb amputees: an epidemiological study. Pain. 2000 Jul;87(1):33-41. doi: 10.1016/S0304-3959(00)00264-5. PMID 10863043
- [Background] Dijkstra PU, Geertzen JH, Stewart R, van der Schans CP. Phantom pain and risk factors: a multivariate analysis. J Pain Symptom Manage. 2002 Dec;24(6):578-85. doi: 10.1016/s0885-3924(02)00538-9. PMID 12551807
- [Background] Richardson C, Glenn S, Nurmikko T, Horgan M. Incidence of phantom phenomena including phantom limb pain 6 months after major lower limb amputation in patients with peripheral vascular disease. Clin J Pain. 2006 May;22(4):353-8. doi: 10.1097/01.ajp.0000177793.01415.bd. PMID 16691088
- [Background] Whyte A, Niven CA. The illusive phantom: does primary care meet patient need following limb loss? Disabil Rehabil. 2004 Jul 22-Aug 5;26(14-15):894-900. doi: 10.1080/09638280410001708904. PMID 15497918
- [Background] Sherman RA, Sherman CJ, Parker L. Chronic phantom and stump pain among American veterans: results of a survey. Pain. 1984 Jan;18(1):83-95. doi: 10.1016/0304-3959(84)90128-3. PMID 6709380
- [Background] Wartan SW, Hamann W, Wedley JR, McColl I. Phantom pain and sensation among British veteran amputees. Br J Anaesth. 1997 Jun;78(6):652-9. doi: 10.1093/bja/78.6.652. PMID 9215014
- [Background] Amir R, Devor M. Ongoing activity in neuroma afferents bearing retrograde sprouts. Brain Res. 1993 Dec 10;630(1-2):283-8. doi: 10.1016/0006-8993(93)90667-c. PMID 8118694
- [Background] Jain N, Florence SL, Kaas JH. Reorganization of Somatosensory Cortex After Nerve and Spinal Cord Injury. News Physiol Sci. 1998 Jun;13:143-149. doi: 10.1152/physiologyonline.1998.13.3.143. PMID 11390778
- [Background] Flor H, Elbert T, Muhlnickel W, Pantev C, Wienbruch C, Taub E. Cortical reorganization and phantom phenomena in congenital and traumatic upper-extremity amputees. Exp Brain Res. 1998 Mar;119(2):205-12. doi: 10.1007/s002210050334. PMID 9535570
- [Background] Chabal C, Jacobson L, Russell LC, Burchiel KJ. Pain responses to perineuromal injection of normal saline, gallamine, and lidocaine in humans. Pain. 1989 Mar;36(3):321-325. doi: 10.1016/0304-3959(89)90091-2. PMID 2710561
- [Background] Parkes CM. Factors determining the persistence of phantom pain in the amputee. J Psychosom Res. 1973 Mar;17(2):97-108. doi: 10.1016/0022-3999(73)90010-x. No abstract available. PMID 4741689
- [Background] Shukla GD, Sahu SC, Tripathi RP, Gupta DK. Phantom limb: a phenomenological study. Br J Psychiatry. 1982 Jul;141:54-8. doi: 10.1192/bjp.141.1.54. PMID 7116073
- [Background] Jensen MP, Turner JA, Romano JM. What is the maximum number of levels needed in pain intensity measurement? Pain. 1994 Sep;58(3):387-392. doi: 10.1016/0304-3959(94)90133-3. PMID 7838588
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Kazis LE, Ren XS, Lee A, Skinner K, Rogers W, Clark J, Miller DR. Health status in VA patients: results from the Veterans Health Study. Am J Med Qual. 1999 Jan-Feb;14(1):28-38. doi: 10.1177/106286069901400105. PMID 10446661
- See also: Southern California Institute for Research and Education Website — http://www.scire-lb.org/